CLINICAL TRIAL: NCT02325843
Title: The Subconjunctival Injection of Human Bone Marrow Mesenchymal Stem Cells for Ocular Corneal Burn: Prospective, Case Series Study
Brief Title: the Treatment of Human Bone Marrow Mesenchymal Stem Cells in Ocular Corneal Burn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, M.D, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014MEKY059
Record Dates: First submitted 2014-12-10; First posted 2014-12-25 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Chemical Burns
MeSH Terms: conditions — Burns, Chemical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- human bone marrow MSC (Experimental): 5×106/0.5ml MSC was injected subconjunctival at the inferior fornix.If persistent epithelial defect was noted thereafter, a second AMT and MSC injection was performed.
  Interventions: Other: human bone marrow MSC

INTERVENTIONS:
Other: human bone marrow MSC — The arms of active comparator :human bone marrow MSC subconjunctival injection once time. If persistent epithelial defect was noted thereafter, a second MSC injection was performed.

SUMMARY:
Ocular chemical burn is one of the cause of vision loss in our country, and there are no satisfactory treatment. Human bone marrow mesenchymal stem cells (MSC) have the biological characteristics of self-renewal, immune regulation, multidirectional differentiation and tissue repair. Our preliminary research showed that in corneal alkali injury rats, the MSC can accelerated the cornea repair, inhibited angiogenesis. The aim of this study is to access the efficacy and safety of mesenchymal stem cell in the treatment of corneal burn in human.

DETAILED DESCRIPTION:
Corneal burn is a ocular damage disease included chemically burned and thermally burned. Surgery of corneal transplantation，amniotic membrane transplantation are some of effective,however,these therapy are expensive and the transplantation resources are limited. To arrest the inflammatory phase, several types of immunosuppressive treatments have been investigated. Corticosteroids also is important, however, long time usage of corticosteroids often cause severe side-effects. Human bone marrow mesenchymal stem cells (MSC) have the biological characteristics of self -renewal, immune regulation, multidirectional differentiation and tissue repair. Our preliminary research showed that in corneal alkali injury rats, the MSC can accelerated the cornea repair, inhibited angiogenesis. Many animal research also revealed that MSC have effect on the ocular alkali burned. And subconjunctivity injection is efficient, the clinical study of MSC on treating other disease have been developed rapidly recently, in further ,the outcome are encouraging, and no side-effect related MSC was reported, MSC can come from bone marrow, Umbilical cord blood，Adipose tissue and so on, but bone marrow MSC is mostly common used. The investigators propose to assess the efficacy and safety of human bone marrow mesenchymal stem cell in the treatment of corneal burn in human.

ELIGIBILITY:
Inclusion Criteria:

1. must be ocular burns including chemically burned or the thermally burned
2. the severity degree should above the Ⅳ degree,including the Ⅳ degree(according the classification of Dua standard,2001)
3. the subjects are willing to accept this research,and promise to coordinate with the researchers during the follow up period
4. the subjects should abide by the laws and rules of the study.
5. the incident time should be within 2 weeks -

Exclusion Criteria:

1. the visual acuity is blind in any of the eye
2. have corneal perforation or have the corneal perforation tendency
3. have been accepted surgury on eyeball after trauma
4. IOP≥25mmHg even after antiglaucoma
5. have the history of other corneal diseaze or surgury
6. have the history of radiotherapy or surgury in the eyeball
7. associated with corneal ulcer or endoophthalmitis
8. uncontrolled hypertension(≥150/95mmHg)
9. abnormal liver and renal function
10. the pregancy women -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events by subconjunctival injection of BMMSCs | 6 months
  Record the adverse events, including topical complications such as ocular infection, conjunctival necrosis at the injection site, retinal artery occlusion, and systemic complications such as fever, urticaria, hemolysis, hypotension, renal and liver dysfunction, tumor formation, and/or abnormalities in complete blood counts.

SECONDARY OUTCOMES:
Incidence of corneal perforation rate after subconjunctival injection of BMMSCs | 6 months
  the number of corneal perforation eyes/total eyes
Time of corneal epithelialization | 6 month
  record the time when cornea finish epithelialization
Visual acuity | 6 month
  Use the visual chart to record the decimal visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Liang Dan, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Le Blanc K, Mougiakakos D. Multipotent mesenchymal stromal cells and the innate immune system. Nat Rev Immunol. 2012 Apr 25;12(5):383-96. doi: 10.1038/nri3209. PMID 22531326
- [Background] Gao XH, Roberts A. The left triangular ligament of the liver and the structures in its free edge (appendix fibrosa hepatis) in Chinese and Canadian cadavers. Am Surg. 1986 May;52(5):246-52. PMID 3706914
- [Result] Hargraves MM. Discovery of the LE cell and its morphology. Mayo Clin Proc. 1969 Sep;44(9):579-99. No abstract available. PMID 4186059
- See also: Multipotent mesenchymal stromal cells and the innate immune system — http://www.ncbi.nlm.nih.gov/pubmed/22531326
- See also: Immunoregulatory properties of clinical grade mesenchymal stromal cells: evidence, uncertainties, and clinical application — http://www.ncbi.nlm.nih.gov/pubmed/23742637
- See also: Modulation of the Early Inflammatory Microenvironment in the Alkali-Burned Eye by Systemically Administered Interferon-gamma-Treated Mesenchymal Stromal Cells — http://www.ncbi.nlm.nih.gov/pubmed/24849741